CLINICAL TRIAL: NCT01268774
Title: Preventive Treatment of VETD in Patients With Multiple Myeloma Receiving Chemotherapy With Thalidomide or Lenalinomide
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: Melisse study
Record Dates: First submitted 2010-12-30; First posted 2010-12-31 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with multiple myeloma have seen their survival rate strongly improved with the use of new anti angiogenic agents. Among them, the new chemotherapy with thalidomide or lenalinomide are frequently successfully suggested in therapeutic protocol such as MPT however they can strongly increase the risk of venous thrombo embolic disease (DVT and PTE) up to 20%. In these conditions, a prevention of this risk can be proposed by physician with either low molecular weight heparin (LMWH) anticoagulants or antiplatelets agents. Pending the new recommendations on the management of VTED, the purpose of this study is to describe in real life conditions the management by oncologists of the thrombo embolic risk for such patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma receiving a chemotherapy protocol including thalidomide or lenalidomide

Exclusion Criteria:

* Patients involved in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patinets with multiple myeloma treated with thalidomide or lenalidomide
Sampling Method: Non-Probability Sample
Enrollment: 529 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Disease history and VETD risk factors. Chemotherapy protocol for multiple myeloma. Therapeutic used for VETD prevention (LWMH, anticoagulants, antiplatelets or none) | 4 months

SECONDARY OUTCOMES:
PE and DVT rate at 4 months and one year. Bleedings and all relevant SAE and AE at 4 months and one year. | 12 months